CLINICAL TRIAL: NCT00099710
Title: A Phase II, Double-Blind, Placebo-Controlled Study of the Safety and Tolerability of Two Doses of Curcumin C3 Complex Versus Placebo in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Curcumin in Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Douglas French Foundation (Other)
Collaborators: Institute for the Study of Aging (ISOA) (Other)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0065
Record Dates: First submitted 2004-12-17; First posted 2004-12-20 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Alzheimer's Disease
Keywords: Curcumin; Turmeric; Curry; NSAID; anti-inflammatory; Cholesterol; anti-oxidant
MeSH Terms: conditions — Alzheimer Disease

INTERVENTIONS:
Dietary Supplement: Curcumin C3 Complex

SUMMARY:
The purpose of this study is to examine the safety and tolerability of curcumin, and to determine its effect on patients with mild to moderate Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
Curcumin, a yellow substance found in the spice Turmeric, has antioxidant, non-steroidal anti-inflammatory (NSAID), and cholesterol-lowering properties, all of which make it a good candidate in the prevention and treatment of AD. The study will examine the safety and tolerability of 2 different doses of curcumin C3 complex. Blood and cerebrospinal fluid (CSF) tests will be used to examine how the curcumin is absorbed in the body, and whether it has an effect on inflammation, oxidative damage, and cholesterol levels. Participants will also be tested to determine the potential effect of curcumin on cognition, behavior, and daily function in patients with mild to moderate AD.

Participants will be randomly assigned to receive one of two doses of curcumin, or a placebo, for the initial 6 months of the trial. For the final 6 months, those receiving a placebo will be switched to one of the two doses of the drug. The 33 participants will make 7 visits to the study site over a 12-month period. These visits may include a physical and neurological examination, routine laboratory tests, lumbar puncture, and neuropsychological (mood and memory) evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 50 years old
* Diagnosis of probable AD
* No history of significant psychiatric or non-AD neurological disease
* Proficient in English to be able to perform cognitive testing
* Caregiver available to monitor and administer medication and to accompany patient to every clinical visit
* On stable doses of cholinesterase inhibitors and memantine (Alzheimer's medications) for 3 months prior to enrollment
* On stable doses of all other allowed medications for at least one month prior to starting the study medication

Exclusion Criteria:

* Current or recent major psychiatric illness (i.e. bipolar disorder, schizophrenia)
* Significant, uncontrolled systemic illness (i.e. chronic renal failure, chronic liver disease, poorly controlled diabetes, or poorly controlled congestive heart failure)
* Recent history of gastrointestinal bleeding or ulceration
* Alcoholism or substance abuse within the past year
* Familial, autosomal dominant Alzheimer's disease due to a mutation in a known gene (Presenilin-1, Presenilin-2, or Amyloid Precursor Protein)
* NSAIDs (e.g. ibuprofen, naproxen, etc.) taken on a regular basis (more than 3 times per week)
* Aspirin at doses more than 325 mg per day
* Coumadin, heparin, other anticoagulants
* Antioxidants or other supplements including gingko biloba, coenzyme Q10, alpha-lipoic acid
* Vitamin E at doses more than 2,000 IU per day
* Vitamin C at doses more than 500 mg per day

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2003-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Side effect checklist

SECONDARY OUTCOMES:
Oxidative damage
Inflammation/gliosis
A-beta levels
Tau levels
Total plasma cholesterol, LDL and HDL; ApoE
Plasma curcumin and metabolites
Cognitive and behavioral measures

CONTACTS AND LOCATIONS:
Overall Officials: John Ringman, MD, Study Director — University of California, Los Angeles
Locations (1):
- UCLA Medical Center, Westwood, Los Angeles, California, United States

REFERENCES:
- [Background] Chandra V, Pandav R, Dodge HH, Johnston JM, Belle SH, DeKosky ST, Ganguli M. Incidence of Alzheimer's disease in a rural community in India: the Indo-US study. Neurology. 2001 Sep 25;57(6):985-9. doi: 10.1212/wnl.57.6.985. PMID 11571321
- [Background] Lim GP, Chu T, Yang F, Beech W, Frautschy SA, Cole GM. The curry spice curcumin reduces oxidative damage and amyloid pathology in an Alzheimer transgenic mouse. J Neurosci. 2001 Nov 1;21(21):8370-7. doi: 10.1523/JNEUROSCI.21-21-08370.2001. PMID 11606625
- [Background] Yang F, Lim GP, Begum AN, Ubeda OJ, Simmons MR, Ambegaokar SS, Chen PP, Kayed R, Glabe CG, Frautschy SA, Cole GM. Curcumin inhibits formation of amyloid beta oligomers and fibrils, binds plaques, and reduces amyloid in vivo. J Biol Chem. 2005 Feb 18;280(7):5892-901. doi: 10.1074/jbc.M404751200. Epub 2004 Dec 7. PMID 15590663
- [Derived] Ringman JM, Frautschy SA, Teng E, Begum AN, Bardens J, Beigi M, Gylys KH, Badmaev V, Heath DD, Apostolova LG, Porter V, Vanek Z, Marshall GA, Hellemann G, Sugar C, Masterman DL, Montine TJ, Cummings JL, Cole GM. Oral curcumin for Alzheimer's disease: tolerability and efficacy in a 24-week randomized, double blind, placebo-controlled study. Alzheimers Res Ther. 2012 Oct 29;4(5):43. doi: 10.1186/alzrt146. eCollection 2012. PMID 23107780